CLINICAL TRIAL: NCT02967965
Title: CARIM Cohort (CARdioprotection in Myocardial Infarction)
Brief Title: CARdioprotection in Myocardial Infarction
Acronym: CARIM
Status: Active, not recruiting | Type: Observational
Sponsor: EZUS-LYON 1 (Other)
Responsible Party: Sponsor
Other Study IDs: CARIM
Record Dates: First submitted 2016-11-10; First posted 2016-11-18 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Myocardial Infarct
Keywords: clinical confounders; myocardial infarction size; determinants of myocardial infarct injury
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — J2-4: 63 mL (3 dry tubes ; 2 citrate tubes and 4 tubes with EDTA, with 2 for DNA isolation) M6: 28 mL (2 dry tube, 1 citrate tube and 1 tube with EDTA) M12: 21 mL (1 dry tube, 1 citrate tube and 1 tube with EDTA) Optional: In centers adequately equipped for management of blood samples in the catheterization laboratory, blood samples will be also taken at JO, before and 4 hours after reperfusion (14 ml each: 1 dry tube and 1 tube with EDTA) after obtention of the agreement of the patient to be included in the cohort CARIM.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Clinical Evaluation, Coronarography, Imagery by MRI, Echocardiography and Biological samples will be collected for each patient.
  Interventions: Other: Imagery

INTERVENTIONS:
Other: Imagery — MRI at year 3
  Other Names: MRI

SUMMARY:
CARIM is a prospective cohort of 2,000 patients with a first myocardial infarction and undergoing reperfusion therapy. Therefore, male and female patients older than 18 years and younger than 90 years with onset of chest pain of less than 12 hours who need a primary percutaneous coronary intervention (PCI) for a ST elevation segment MI (STEMI) will be recruited.

DETAILED DESCRIPTION:
In the setting of research in ischemic cardiomyopathy, the CARIM cohort aims to meet the expectation and strategy of Aviesan (Alliance nationale pour les sciences de la VIE et de la SANté) since it will address the underlying pathophysiology of the determinants of MI injury and its impact on follow-up, in addition with the potential confounding clinical and biological factors. Therefore, CARIM cohort will offer a great opportunity of describing the interactions between myocardial infarction and surrounding environment (clinical, social and professional). This cohort will use complementary state of the art approaches (cardiac imaging including Cardiovascular Magnetic Resonance and echocardiography, biomarkers, proteomic, genetic and pharmacogenetics) with strong interactions between the different partners. Therefore CARIM cohort should help to obtain a modeling of the determinants of the MI size.

The investigators expect that CARIM cohort will provide new imaging or biological markers that may bring early information regarding the severity of lethal reperfusion injury.

By optimizing the knowledge on infarct injury in addition with a 5-year clinical and echographic follow-up, this cohort will better stratify the prognosis after MI and will therefore give new insights in identifying patients at higher risk of left ventricular remodeling and subsequent heart failure. It will therefore help and emphasize prevention messages and patients' education. The aim is to translate this information directly into patient care by using the science generated by this project to develop new management guidelines and novel clinical tools (confounder-annotated database, imaging and biological biomarkers). This cohort may have additional impact in patient care by adapting the treatment to patient-related confounders (age, diabetes...), genetic polymorphisms and thus personalizing health care to individuals.

3.2 MAIN OBJECTIVE

The investigators main objective is to create a prospective cohort of 2,000 patients (CARIM cohort) with a first myocardial infarction and undergoing reperfusion therapy in order to evaluate the impact of patient-related confounders on myocardial infarct size and LRI in order to further design a modeling of myocardial infarct size.

For this purpose, CARIM cohort will be associated with the creation of a non-invasive cardiac imaging data-bank (MRI and echocardiography) in addition with a large bio-bank relying on existing biological certified platforms (i.e. BRC network).

This cohort will provide a population of first acute MI, optimally characterized in terms of comprehensive clinical and angiography phenotype, specifically characterized by CMR in terms of infarct size and LRI and by echocardiography in terms of myocardial regional function and left ventricular remodeling.

3.3 SECONDARY OBJECTIVES

1. Evaluate the specific impact of myocardial infarct injury on myocardial regional function and left ventricular remodeling (defined by an increase in LV end-diastolic volume > 20% between week 1 and month 12 post-MI by echocardiography).
2. Evaluate the power of the myocardial infarct injury in predicting cardiovascular events (rehospitalizations, reinfarction, occurrence of HF, transplantation, arrhythmias, death) in a 5-year patient follow-up.
3. Test the value of established or newly identified plasma/serum biomarkers to identify LRI and to predict post-MI LV remodeling and progression towards CHF during a 5 year follow-up.
4. This cohort aims ultimately at defining the profile of the MI patient population to be used for future trials implementing new protective interventions targeting LRI.

ELIGIBILITY:
Inclusion Criteria:

Any patient hospitalized in the cardiology department of the participating centers

* Who have signed the Informed Consent Form.
* Patient having health insurance.
* Requiring PCI for reperfusion.
* With a diagnosis of a first MI.
* With ST segment elevation and/or Q wave at admission.
* With troponin elevation.
* Seen within the first 12 hours after symptom onset.
* Aged between 18 and 90 years.

Exclusion Criteria:

* Refusal of the patient.
* In case of poor echogenicity, the participation of the patient will be stopped.
* Patient with diagnosis of previous MI, or hypertrophic or dilated cardiomyopathy, or significant valvular heart disease, or chronic atrial fibrillation, or pace maker or any permanent implanted device susceptible to interfere with LV remodeling.
* Patient with preexisting heart failure.
* Patient with any previous cardiac surgery.
* Patient with previous chemotherapy susceptible to induce LV remodeling (anthracyclines).
* Patient with an associated short-time life-threatening disease.
* Pregnant or breast-feeding patient.
* Contra-indication to MRI (claustrophobia, pacemaker or any other metallic implants, creatinin clearance < 30mL/min/1.73m2 MDRD).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CARIM is a prospective cohort of 2,000 patients with a first myocardial infarction and undergoing reperfusion therapy. Therefore, male and female patients older than 18 years and younger than 90 years with onset of chest pain of less than 12 hours who need a primary percutaneous coronary intervention (PCI) for a ST elevation segment MI (STEMI) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-11-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Determinants of myocardial infarct injury | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve DERUMEAUX, Professor, Principal Investigator — APHP
Locations (2):
- France (2):
  - CHRU de Tours, Tours, Indre Et Loire
  - Hôpital Mondor, Créteil, Rhône

IPD SHARING:
Plan to Share IPD: No